CLINICAL TRIAL: NCT04072575
Title: Single-arm, Open-label Extension to a Double-blind, Randomized, Active-controlled, Parallel-group Study of Paliperidone Palmitate 6-Month Formulation
Brief Title: A Study of Paliperidone Palmitate 6-Month Formulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108605; R092670PSY3016 (Other: Janssen Research & Development, LLC); 2018-004532-30 (EudraCT Number)
Record Dates: First submitted 2019-08-16; First posted 2019-08-28 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Paliperidone Palmitate 6 month(PP6M) (Experimental): Participants who enter the this open-label extension study immediately after completing Double-blind Phase Study R092670PSY3015 (previous study) will receive Paliperidone Palmitate 6 month (PP6M) intramuscular (IM) injections, dose will be selected based on the unblinded dose level ("moderate" or "higher") that the participant received during previous study. Participants in the "moderate" dose level will receive PP6M Dose 1 and "higher" dose level will receive PP6M Dose 2 during the open-label extension. The PP6M dose level may be adjusted (to Dose 1 or Dose 2) for every 6 month at Visits 3, 5, and 7, based on clinical judgment. Participants who enter this open-label extension study later (up to 3 months after they complete previous study) and were on a moderate or higher dose of PP3M (350 or 525 mg eq.) or PP1M (100 or 150 mg eq.) will receive initial dose of PP6M IM injection (Dose 1 or Dose 2) for every 6 months.
  Interventions: Drug: PP6M injection Dose 1; Drug: PP6M injection Dose 2

INTERVENTIONS:
Drug: PP6M injection Dose 1 — Participants will receive Dose 1 PP6M intramuscular (IM) injection at Visit 1 (Day) then once every 6 month up to 24 months.
  Other Names: R092670
Drug: PP6M injection Dose 2 — Participants will receive Dose 2 PP6M IM injection at Visit 1 (Day) then once every 6 month up to 24 months.
  Other Names: R092670

SUMMARY:
The main purpose of this study is to assess the long-term safety and tolerability of paliperidone 6-month PP6M (Dose 1 or Dose 2 [milligram] mg eq.) and to provide access to PP6M in participants with schizophrenia completing the R092670PSY3015 study without relapse.

ELIGIBILITY:
Inclusion Criteria:

* Completed the Double-blind Phase of Study R092670PSY3015 without relapse and continue to be willing to be treated with paliperidone palmitate 6 month injection (PP6M)
* Must, in the opinion of the investigator, be able to continue treatment at the same dose level (moderate or higher dose) as used during the Double-blind Phase of Study R092670PSY3015 at the time of screening for this study
* A woman of childbearing potential: a) Must have a negative pregnancy test on Day 1; b) Use contraception consistent with local regulations. A man must agree that during the study and for a minimum 12 months after receiving the last dose of the study intervention: a) His female partner(s) will use highly effective method pf contraception
* Sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study; and must be able to provide his or her own consent (that is, consent cannot be provided by a legal representative of the participant)
* In the opinion of the investigator, the patient would be able to participate for the duration of this study

Exclusion Criteria:

* Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Completed R092670PSY3015 while presenting adverse events deemed clinically relevant by the investigator, and which may interfere with safety and well-being of the participant
* If a man, has plans to father a child while enrolled in this study or within 12 months after the last dose of study intervention. Must not, if a woman, have plans to become pregnant while enrolled in this study or within 12 months after the last dose of study intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (30):
- Argentina (6):
  - Fundacion para el Estudio y Tratamiento de las Enfermedades Mentales, Buenos Aires
  - CEN Consultorios Especializados en Neurociencias, Córdoba
  - Sanatorio Prof. Leon S. Morra, Córdoba
  - INSA Instituto de Neurociencias San Agustín, La Plata
  - Clinica Privada de Salud Mental Santa Teresa de Ávila, La Plata
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
- Queen Mary Hospital, Hong Kong, Hong Kong
- Italy (3):
  - Dipartimento di Salute Mentale, Lecce
  - Seconda Universita degli Studi di Napoli - Azienda Ospedaliera Universitaria, Napoli
  - Universita degli Studi di Roma 'La Sapienza' - Azienda Ospedaliera Sant Andrea, Roma
- Poland (7):
  - Mlynowamed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk, Bialystok
  - Zespol Opieki Zdrowotnej w Chelmnie, Chełmno
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Specjalistyczna Praktyka Lekarska Piotr Zalitacz, Gorlice
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Centrum Medyczne Luxmed Sp z o o, Lublin
  - Poradnia Zdrowia Psychicznego 'Syntonia' w Pruszczu Gdanskim, Pruszcz Gdański
- Russia (5):
  - Nizny Novgorod clinical psychiatric hospital 1, Nizny Novgorod
  - SHI 'Saratov City Clinical Hospital 2 n.a V.I. Razumovsky, Saratov
  - Saratov Regional Psychiatric hospital named after St. Sofia, Saratov
  - Research Institute of Mental Health, Tomsk
  - Sverdlovsk Regional Clinical Psychiatric Hospital, Yekaterinburg
- Ukraine (8):
  - MNCE of Kyiv RC Regional Psychiatric and Narcological Medical Association, Hlevakha
  - Mnpe of Kharkiv Regional Council 'Regional Clinical Psychiatric Hospital #3', Kharkiv
  - CNPE'Kherson Regional Institution of Mental Care'of Kherson Regional Council, Kherson
  - Mnpe of Lviv Regional Council 'Lviv Regional Clinical Psycho-Neurological Dispensary', Lviv
  - CNCE of the Lviv Regional Council 'Lviv Regional Clinical Psychiatric Hospital', Lviv
  - CNCE Odesa regional psychiatric hospital #2 Odesa regional council, Oleksandrivka
  - CNCE 'Cherkasy Regional Psychiatric Hospital of Cherkasy Regional Council', Smila
  - CNCE 'Vinnytsya RC Psychoneurological Hospital n.a. O.I. Yushchenko Vinnytsya RC', Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] LaRoche JK, Lanier J, Alvarenga R, Collins M, Costelloe T, Chiau A, Whetherly H, De Soete W, Faludi J, Rens K. Climate footprint of industry-sponsored in-human clinical trials: life cycle assessments of clinical trials spanning multiple phases and disease areas. BMJ Open. 2025 Feb 19;15(2):e085364. doi: 10.1136/bmjopen-2024-085364. PMID 39971605
- [Derived] Turkoz I, Daskiran M, Siddiqui U, Knight RK, Johnston KL, Correll CU. Relapse Rates With Paliperidone Palmitate in Adult Patients With Schizophrenia: Results for the 6-Month Formulation From an Open-label Extension Study Compared to Real-World Data for the 1-Month and 3-Month Formulations. Int J Neuropsychopharmacol. 2024 Feb 1;27(2):pyad067. doi: 10.1093/ijnp/pyad067. PMID 38300235
- [Derived] Najarian D, Turkoz I, Knight RK, Galderisi S, Lamaison HF, Zalitacz P, Aravind S, Richarz U. Long-Term Efficacy and Safety of Paliperidone 6-Month Formulation: An Open-Label 2-Year Extension of a 1-Year Double-Blind Study in Adult Participants With Schizophrenia. Int J Neuropsychopharmacol. 2023 Aug 29;26(8):537-544. doi: 10.1093/ijnp/pyad028. PMID 37480362

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.: Participants who completed the 12-month double-blind (DB) phase of study R092670PSY3015 (NCT03345342) without a relapse, were enrolled in this open-label extension (OLE) study and received intramuscular (IM) injections of PP6M 700 (if received moderate dose previously) or 1000 milligrams equivalent (mg eq.) (if received higher dose previously) on Day 1. On Days 183, 365, and 547, flexible dosings were permitted to increase PP6M 700 mg eq. to 1000 mg eq. or decrease 1000 mg eq. to 700 mg eq. as per investigator's judgement.
Period: Overall Study
Arm/Group | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.
Started | 178
Completed | 154
Not Completed | 24
Not completed — Physician Decision | 1
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 14
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48
  Not Hispanic or Latino | 130
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 176
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse
Description: Number of participants with relapse were reported. Relapse is defined as one or more of the following: a) Psychiatric hospitalization for schizophrenia (involuntary or voluntary admission to a psychiatric hospital for decompensation of the participant's schizophrenic symptoms); b) Emergency Department/Room/Ward visit due to a worsening of the participant's symptoms of schizophrenia, but a psychiatric hospitalization does not occur; c) The participant inflicts deliberate self-injury or exhibits violent behaviour resulting in suicide, clinically significant injury to him/herself or another person, or significant property damage; d) The participant has suicidal or homicidal ideation and aggressive behaviour that is clinically significant (in frequency and severity) in the investigator's judgment.
Time Frame: Up to Day 730
Population: The intent-to-treat (ITT) analysis population included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.
Number analyzed (Participants) | 178
Participants | 7

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. TEAEs are those events if they started after administration of the first dose and until 183 days after the last dose of study medication.
Time Frame: Up to Day 730
Population: The safety analysis population included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.
Number analyzed (Participants) | 178
Participants | 111

3. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Scale Score
Description: Change from baseline in CGI-S scale score was reported. CGI-S is defined as clinician-rated scale that assesses the severity of mental illness on a scale of 0 to 7. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating according to:1: normal, not at all ill; 2: borderline mentally ill; 3: mildly ill; 4: moderately ill; 5: markedly ill; 6: severely ill; 7: among the most extremely ill participants. A higher score implies a more severe condition.
Time Frame: Baseline up to Day 730
Population: The ITT analysis population included all participants who received at least 1 dose of study drug in this study. Here, 'N' (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.
Number analyzed (Participants) | 176
Units on a scale | 0.0 (0.51) [lower limit 0.51]

4. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) Scale Score
Description: Change from baseline in PSP scale score was reported. The PSP scale assesses degree of a participant's dysfunction within 4 domains of behavior: 1) socially useful activities, 2) personal and social relationships, 3) self-care, and 4) disturbing and aggressive behavior. Each domain was assessed on a 6-point scale, from 1 (absent) to 6 (very severe) (1 = absent, 2 = mild, 3 = manifest, 4 = marked, 5 = severe, and 6 = very severe). PSP total score was calculated as sum of all the domain scores and ranges from 1 to 100. Participants with score of 71 to 100 had mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision. Higher score indicates better performance.
Time Frame: Baseline up to Day 730
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.
Number analyzed (Participants) | 173
Units on a scale | 0.5 (7.47) [lower limit 7.47]

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: Change from baseline in PANSS total score were reported. The neuropsychiatric symptoms of schizophrenia were assessed using the 30-item PANSS scale, which provides a total score (sum of the scores for all 30 items) and scores for 3 subscales: the 7-item positive-symptom (P) subscale, the 7-item negative-symptom (N) subscale, and the 16-item general-psychopathology symptom (G) subscale. Each item is rated on a scale of 1 (absent) to 7 (extreme). The PANSS total score ranges from 30 (absent disease)-210 (more severe neuropsychiatric symptoms of schizophrenia).
Time Frame: Baseline up to Day 730
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.
Number analyzed (Participants) | 173
Units on scale | 0.7 (8.22) [lower limit 8.22]

ADVERSE EVENTS:
Time Frame: Up to Day 730
Description: The safety analysis population included all participants who received at least 1 dose of study drug in this study.
Arm/Group | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq.
All-Cause Mortality (participants affected / at risk) | 0/178
Serious Adverse Events (participants affected / at risk) | 8/178
Other Adverse Events (participants affected / at risk) | 68/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq. (N=178)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hallucination, Auditory (Psychiatric disorders) | 1 (1)
Psychiatric Symptom (Psychiatric disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 4 (4)
Nephrotic Syndrome (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Paliperidone Palmitate 6-month (PP6M) 700 or 1000 mg eq. (N=178)
Hyperprolactinaemia (Endocrine disorders) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 11 (12)
Nasopharyngitis (Infections and infestations) | 9 (11)
Blood Prolactin Increased (Investigations) | 19 (19)
Weight Increased (Investigations) | 9 (9)
Headache (Nervous system disorders) | 24 (30)

LIMITATIONS AND CAVEATS:
The sponsor identified that the study did not include a control arm reference group. The coronavirus disease-2019 (COVID-19) pandemic placed some restrictions on study face-to-face visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT04072575/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT04072575/SAP_001.pdf